CLINICAL TRIAL: NCT00853723
Title: Comparison of 3 Month PTHrP(1-36) and PTH(1-34) on Post-Menopausal Osteoporosis
Brief Title: Comparison Study of PTHrP and PTH to Treat Osteoporosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Mara Horwitz, Associate Professor, University of Pittsburgh School of Medicine, University of Pittsburgh
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: PRO08100148; R01DK051081 (NIH)
Record Dates: First submitted 2009-02-27; First posted 2009-03-02 (Estimated); Results first posted 2016-02-24 (Estimated); Last update posted 2016-03-24 (Estimated); Status verified 2016-02

CONDITIONS: Osteoporosis
Keywords: osteoporosis; post-menopausal; bone anabolic agents
MeSH Terms: conditions — Osteoporosis | interventions — parathyroid hormone-related peptide (1-36); Parathyroid Hormone-Related Protein; Parathyroid Hormone; Teriparatide

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- PTHrP 400 mcg/day (Experimental): Post-menopausal women with osteoporosis will subcutaneously administer PTHrP 400 micrograms daily for three months.
  Interventions: Drug: Parathyroid hormone related protein (1-36)
- PTHrP 600 mcg/day (Experimental): Post-menopausal women with osteoporosis will subcutaneously administer PTHrP 600 micrograms daily for three months.
  Interventions: Drug: Parathyroid hormone related protein(1-36)
- PTH 20 mcg/day (Active Comparator): Post-menopausal women with osteoporosis will subcutaneously administer the FDA approved dose of PTH 20 micrograms daily for three months.
  Interventions: Drug: Parathyroid hormone (1-34)

INTERVENTIONS:
Drug: Parathyroid hormone related protein (1-36) — PTHrP (1-36) 400 micrograms / day administered subcutaneously for 3 months
  Other Names: PTHrP (1-36); PTHrP
  Arms: PTHrP 400 mcg/day
Drug: Parathyroid hormone related protein(1-36) — PTHrP(1-36)600 micrograms subcutaneously administered daily for 3 months
  Other Names: PTHrP (1-36); PTHrP
  Arms: PTHrP 600 mcg/day
Drug: Parathyroid hormone (1-34) — PTH(1-34)20 micrograms subcutaneously administered daily for 3 months
  Other Names: PTH(1-34); Teriparatide (brand name: Forteo)
  Arms: PTH 20 mcg/day

SUMMARY:
This is a three month comparison trial of standard dose parathyroid hormone (PTH) (1-34) and two different doses of Parathyroid Hormone-related Protein (PTHrP) (1-36). The investigators want to to demonstrate that daily subcutaneous injection of PTHrP (1-36) in postmenopausal women with osteoporosis stimulates bone formation to the same or greater degree than PTH (1-34) but with less bone resorption.

DETAILED DESCRIPTION:
Osteoporosis is a metabolic bone disease characterized by low bone mass and structural deterioration of bone tissue. It results from failure of osteoblasts to form sufficient new bone, from an excessive rate of osteoclastic bone resorption, or from the combination of both processes. The resultant bone fragility leads to an increased susceptibility to fractures, especially of the hip, spine and wrist. There is an increased mortality rate following both hip and vertebral fractures, and the presence of one fracture is a potent risk factor for future fractures. This leads to a decline in the quality of life and an associated loss of independence among the millions of individuals in the United States and worldwide afflicted with the disease. There is an additional population at an increased risk for fractures due to a less severe loss of bone mass, known as osteopenia (1). Already ten million individuals in the United States are estimated to have the disease and thirty four million more are at increased risk due to low bone mass (1).

Approved pharmacological treatments for postmenopausal osteoporosis include two classes of drugs: the antiresorptive and the anabolics (2). The antiresorptive include estrogen, calcitonin, selective estrogen receptor modulators, and bisphosphonates. The antiresorptive medications prevent bone loss by inhibiting both osteoclastic bone resorption and formation, by slowing bone turnover, and by allowing for increased mineralization of osteoid (2). The increase in bone mineral density from the antiresorptive agents is generally reported to be in the range of 2-8% over 1-7 years (3-7).

There is only one anabolic agent that is presently approved by the FDA for treatment for osteoporosis: parathyroid hormone, PTH (1-34), or teriparatide. PTH(1-34) was approved by the FDA in 2002 and it acts by increasing bone density by stimulating the PTH-1 receptor. This induces an increase in osteoblast mediated bone formation and osteoclast mediated bone resorption. Daily subcutaneous PTH is anabolic as there is stimulation of bone formation to a greater extent than bone resorption. The overall net result of biosynthetic PTH (1-34) is an increase in bone mineral density and a decrease in fractures (8). Daily PTH(1-34) treatment has been shown to effectively reduce the risk of both vertebral and nonvertebral fractures. Measurements of bone mineral density (BMD) of the lumbar spine (LS) resulted in an increase in bone density of 9 percent when compared to placebo (9). A daily 20 microgram dose of subcutaneous PTH(1-34) reduced the risk of getting two or more vertebral fractures by 77%, and the risk of at least one moderate or severe fracture was reduced by 90 and 78% respectively (9). Additionally, one vertebral fracture was prevented for every 12 patient years of treatment, and women were 35% less likely to have one or more new nonvertebral fragility fractures (9).

Parathyroid hormone-related protein or PTHrP is a protein peptide that was first isolated in 1987 as the factor responsible for the syndrome of humoral hypercalcemia of malignancy (HHM) (10-14). PTHrP is found in almost every tissue and cell type in the body, and appears to regulate cellular proliferation, survival, and differentiation in normal tissue as well as in malignancies (15-16). As the name implies, PTHrP is similar to PTH. Both peptides bind to the same receptor, PTH-1 R, and activate downstream signaling pathways causing similar post receptor effects (17).

Since PTH is a potent anabolic agent, we hypothesize that PTHrP may act in an anabolic fashion as well. We are seeking to demonstrate in this study that PTHrP acts as an anabolic agent in the treatment of osteoporosis with similar or better efficacy than PTH in respect to bone formation but with less bone resorption and fewer side effects, such as hypercalcemia.

The current studies are a sequel to initial phase 1 trials assessing the efficacy and safety of daily subcutaneous injection of PTHrP on the human skeleton. Previous studies have demonstrated that a single daily injection of ~ 400 mcg/day of PTHrP (1-36) in postmenopausal women on estrogen with osteoporosis led to a 4.7% increase in lumbar spine bone mineral density (BMD) after three months and all subjects were free of hypercalcemia or other adverse effects (18). In contrast with PTH, the doses of PTHrP are much larger, yet well-tolerated, and the increments in spine BMD are large and rapid with some subjects showing increases in spine BMD of 6-8% in as soon as three months in studies done thus far (18). PTHrP appears to selectively stimulate bone formation without stimulating bone resorption (18). This exciting observation may point towards PTHrP being a pure skeletal anabolic agent (21). Preliminary data analysis from a more recent three week dose escalation trial indicates demonstrates that the dose of 500 mcg/day of PTHrP causes 38% increase in P1NP and a 20% decrease in CTX indicating far greater bone formation than bone resorption with no hypercalcemia. At 625 mcg/day there were similar increases in P1NP with hypercalcemia in only 10% of subjects and hypercalcuria in 20%. In contrast in subjects receiving 750 mcg/day 50% developed hypercalcemia requiring early termination. The P1NP and CTX data from the three week dose escalation trial was used for both determining dose and sample size calculations for this study.

ELIGIBILITY:
Inclusion Criteria:

* 45 - 75 year old Caucasian, Hispanic or Asian women
* one year post-menopausal if older than 50 years
* three years post-menopausal if between the ages of 45 - 50 years
* body mass index less than or equal to 30
* T-scores on screening Dual X-Ray Absorbiometry (DXA) scan between - 2.0 to - 4.5 of lumbar spine or hip
* have at lease two spinal vertebrae evaluable by DXA analysis

Exclusion Criteria:

* bisphosphonate therapy within the last two years
* estrogen replacement hormones or SERMS within last one year
* no more than one week of PTHrP, PTH, or an analog of PTH within the last year
* an atraumatic bone fracture within the last 6 months
* significant or active diseases of any organ system
* history of malignancy
* anemia with a hematocrit less than 34%
* significant drug or alcohol abuse
* having received any investigational drug within the last 90 days
* taking any medication that may interfere with skeletal metabolism, such as phenobarbital, dilantin, glucocorticoids, and hydrochlorathiazide
* abnormal screening labs including serum Ca greater than 10.5 g/dl, 25 hydroxy vitamin D less than 20 ng/ml or PTH greater than 65 pg/ml
* African-Americans for this particular study - although future studies are planned

Ages: 45 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2009-05; Primary Completion 2012-02 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mara J Horwitz, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC Clinical & Translational Research Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] http://www.nof.org/osteoporosis/diseasefacts.htm. Accessed August 22, 2008
- [Background] Black DM, Bouxsein ML, Palermo L, McGowan JA, Newitt DC, Rosen E, Majumdar S, Rosen CJ; PTH Once-Weekly Research (POWR) Group. Randomized trial of once-weekly parathyroid hormone (1-84) on bone mineral density and remodeling. J Clin Endocrinol Metab. 2008 Jun;93(6):2166-72. doi: 10.1210/jc.2007-2781. Epub 2008 Mar 18. PMID 18349061
- [Background] Effects of hormone therapy on bone mineral density: results from the postmenopausal estrogen/progestin interventions (PEPI) trial. The Writing Group for the PEPI. JAMA. 1996 Nov 6;276(17):1389-96. PMID 8892713
- [Background] Liberman UA, Weiss SR, Broll J, Minne HW, Quan H, Bell NH, Rodriguez-Portales J, Downs RW Jr, Dequeker J, Favus M. Effect of oral alendronate on bone mineral density and the incidence of fractures in postmenopausal osteoporosis. The Alendronate Phase III Osteoporosis Treatment Study Group. N Engl J Med. 1995 Nov 30;333(22):1437-43. doi: 10.1056/NEJM199511303332201. PMID 7477143
- [Background] Delmas PD, Bjarnason NH, Mitlak BH, Ravoux AC, Shah AS, Huster WJ, Draper M, Christiansen C. Effects of raloxifene on bone mineral density, serum cholesterol concentrations, and uterine endometrium in postmenopausal women. N Engl J Med. 1997 Dec 4;337(23):1641-7. doi: 10.1056/NEJM199712043372301. PMID 9385122
- [Background] Chesnut CH 3rd, Silverman S, Andriano K, Genant H, Gimona A, Harris S, Kiel D, LeBoff M, Maricic M, Miller P, Moniz C, Peacock M, Richardson P, Watts N, Baylink D. A randomized trial of nasal spray salmon calcitonin in postmenopausal women with established osteoporosis: the prevent recurrence of osteoporotic fractures study. PROOF Study Group. Am J Med. 2000 Sep;109(4):267-76. doi: 10.1016/s0002-9343(00)00490-3. PMID 10996576
- [Background] Fogelman I, Ribot C, Smith R, Ethgen D, Sod E, Reginster JY. Risedronate reverses bone loss in postmenopausal women with low bone mass: results from a multinational, double-blind, placebo-controlled trial. BMD-MN Study Group. J Clin Endocrinol Metab. 2000 May;85(5):1895-900. doi: 10.1210/jcem.85.5.6603. PMID 10843171
- [Background] Neer RM, Arnaud CD, Zanchetta JR, Prince R, Gaich GA, Reginster JY, Hodsman AB, Eriksen EF, Ish-Shalom S, Genant HK, Wang O, Mitlak BH. Effect of parathyroid hormone (1-34) on fractures and bone mineral density in postmenopausal women with osteoporosis. N Engl J Med. 2001 May 10;344(19):1434-41. doi: 10.1056/NEJM200105103441904. PMID 11346808
- [Background] Stewart AF, Horst R, Deftos LJ, Cadman EC, Lang R, Broadus AE. Biochemical evaluation of patients with cancer-associated hypercalcemia: evidence for humoral and nonhumoral groups. N Engl J Med. 1980 Dec 11;303(24):1377-83. doi: 10.1056/NEJM198012113032401. PMID 6253785
- [Background] Stewart AF, Vignery A, Silverglate A, Ravin ND, LiVolsi V, Broadus AE, Baron R. Quantitative bone histomorphometry in humoral hypercalcemia of malignancy: uncoupling of bone cell activity. J Clin Endocrinol Metab. 1982 Aug;55(2):219-27. doi: 10.1210/jcem-55-2-219. PMID 7085851
- [Background] Strewler GJ. The physiology of parathyroid hormone-related protein. N Engl J Med. 2000 Jan 20;342(3):177-85. doi: 10.1056/NEJM200001203420306. No abstract available. PMID 10639544
- [Background] Broadus AE, Mangin M, Ikeda K, Insogna KL, Weir EC, Burtis WJ, Stewart AF. Humoral hypercalcemia of cancer. Identification of a novel parathyroid hormone-like peptide. N Engl J Med. 1988 Sep 1;319(9):556-63. doi: 10.1056/NEJM198809013190906. No abstract available. PMID 3043221
- [Background] Philbrick WM, Wysolmerski JJ, Galbraith S, Holt E, Orloff JJ, Yang KH, Vasavada RC, Weir EC, Broadus AE, Stewart AF. Defining the roles of parathyroid hormone-related protein in normal physiology. Physiol Rev. 1996 Jan;76(1):127-73. doi: 10.1152/physrev.1996.76.1.127. PMID 8592727
- [Background] Orloff JJ, Reddy D, de Papp AE, Yang KH, Soifer NE, Stewart AF. Parathyroid hormone-related protein as a prohormone: posttranslational processing and receptor interactions. Endocr Rev. 1994 Feb;15(1):40-60. doi: 10.1210/edrv-15-1-40. PMID 8156938
- [Background] Horwitz MJ, Tedesco MB, Sereika SM, Hollis BW, Garcia-Ocana A, Stewart AF. Direct comparison of sustained infusion of human parathyroid hormone-related protein-(1-36) [hPTHrP-(1-36)] versus hPTH-(1-34) on serum calcium, plasma 1,25-dihydroxyvitamin D concentrations, and fractional calcium excretion in healthy human volunteers. J Clin Endocrinol Metab. 2003 Apr;88(4):1603-9. doi: 10.1210/jc.2002-020773. PMID 12679445
- [Background] Horwitz MJ, Tedesco MB, Gundberg C, Garcia-Ocana A, Stewart AF. Short-term, high-dose parathyroid hormone-related protein as a skeletal anabolic agent for the treatment of postmenopausal osteoporosis. J Clin Endocrinol Metab. 2003 Feb;88(2):569-75. doi: 10.1210/jc.2002-021122. PMID 12574182
- [Background] Stewart AF, Cain RL, Burr DB, Jacob D, Turner CH, Hock JM. Six-month daily administration of parathyroid hormone and parathyroid hormone-related protein peptides to adult ovariectomized rats markedly enhances bone mass and biomechanical properties: a comparison of human parathyroid hormone 1-34, parathyroid hormone-related protein 1-36, and SDZ-parathyroid hormone 893. J Bone Miner Res. 2000 Aug;15(8):1517-25. doi: 10.1359/jbmr.2000.15.8.1517. PMID 10934650
- [Background] Dean T, Vilardaga JP, Potts JT Jr, Gardella TJ. Altered selectivity of parathyroid hormone (PTH) and PTH-related protein (PTHrP) for distinct conformations of the PTH/PTHrP receptor. Mol Endocrinol. 2008 Jan;22(1):156-66. doi: 10.1210/me.2007-0274. Epub 2007 Sep 13. PMID 17872377
- [Background] Bisello A, Horwitz MJ, Stewart AF. Parathyroid hormone-related protein: an essential physiological regulator of adult bone mass. Endocrinology. 2004 Aug;145(8):3551-3. doi: 10.1210/en.2004-0509. No abstract available. PMID 15265822
- [Background] Horwitz MJ, Tedesco MB, Sereika SM, Garcia-Ocana A, Bisello A, Hollis BW, Gundberg C, Stewart AF. Safety and tolerability of subcutaneous PTHrP(1-36) in healthy human volunteers: a dose escalation study. Osteoporos Int. 2006 Feb;17(2):225-30. doi: 10.1007/s00198-005-1976-3. Epub 2005 Sep 7. PMID 16151606
- [Background] FORTEO (package insert). Indianapolis, IN: Eli Lilly and Company; 2008.
- [Background] Miller PD, Bilezikian JP, Diaz-Curiel M, Chen P, Marin F, Krege JH, Wong M, Marcus R. Occurrence of hypercalciuria in patients with osteoporosis treated with teriparatide. J Clin Endocrinol Metab. 2007 Sep;92(9):3535-41. doi: 10.1210/jc.2006-2439. Epub 2007 Jul 3. PMID 17609307
- [Background] McClung MR, San Martin J, Miller PD, Civitelli R, Bandeira F, Omizo M, Donley DW, Dalsky GP, Eriksen EF. Opposite bone remodeling effects of teriparatide and alendronate in increasing bone mass. Arch Intern Med. 2005 Aug 8-22;165(15):1762-8. doi: 10.1001/archinte.165.15.1762. PMID 16087825
- [Background] Anastasilakis AD, Goulis DG, Polyzos SA, Gerou S, Koukoulis GN, Efstathiadou Z, Kita M, Avramidis A. Head-to-head comparison of risedronate vs. teriparatide on bone turnover markers in women with postmenopausal osteoporosis: a randomised trial. Int J Clin Pract. 2008 Jun;62(6):919-24. doi: 10.1111/j.1742-1241.2008.01768.x. Epub 2008 Apr 17. PMID 18422590
- [Background] Tashjian AH Jr, Gagel RF. Teriparatide [human PTH(1-34)]: 2.5 years of experience on the use and safety of the drug for the treatment of osteoporosis. J Bone Miner Res. 2006 Mar;21(3):354-65. doi: 10.1359/JBMR.051023. Epub 2005 Nov 11. No abstract available. PMID 16491282
- [Background] Horwitz MJ, Stewart Af. Humoral hypercalcemia of malignancy. In: Favus MF (ed.) Primer on Metabolic Bone Diseases and Disorders of Mineral Metabolism, 5th ed. American Society for Bone and Mineral Research, Washington, DC, USA, pp. 246-250:2003.
- [Background] Lachin JM. Introduction to sample size determination and power analysis for clinical trials. Control Clin Trials. 1981 Jun;2(2):93-113. doi: 10.1016/0197-2456(81)90001-5. PMID 7273794

RESULTS

PARTICIPANT FLOW:
Groups:
- PTHrP 400 mcg/Day: Post-menopausal women with osteoporosis or low bone density will subcutaneously administer Parathyroid hormone related protein (PTHrP) 1-36, 400 micrograms / day for 3 months
- PTHrP 600 mcg/Day: Post-menopausal women with osteoporosis or low bone density will subcutaneously administer Parathyroid hormone related protein (PTHrP) 1-36, 600 micrograms / day for 3 months
- PTH 20 mcg/Day: Post-menopausal women with osteoporosis or low bone density will subcutaneously administer Parathyroid hormone (PTH) 1-34, 20 micrograms / day for 3 months
Period: Overall Study
Arm/Group | PTHrP 400 mcg/Day | PTHrP 600 mcg/Day | PTH 20 mcg/Day
Started | 35 | 35 | 35
Completed | 29 | 28 | 33
Not Completed | 6 | 7 | 2
Not completed — Adverse Event | 3 | 4 | 1
Not completed — Withdrawal by Subject | 2 | 1 | 0
Not completed — Protocol Violation | 1 | 2 | 1

BASELINE CHARACTERISTICS:
Population: Postmenopausal women age 45-75 with osteoporosis or low bone density
Groups:
- Total: Total of all reporting groups
Arm/Group | PTHrP 400 mcg/Day | PTHrP 600 mcg/Day | PTH 20 mcg/Day | Total
Number analyzed (Participants) | 35 | 35 | 35 | 105
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 28 | 25 | 25 | 78
  >=65 years | 7 | 10 | 10 | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.6 (5.22) | 61.2 (5.10) | 62.4 (5.26) | 61.4 (5.20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 35 | 35 | 105
  Male | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 35 | 35 | 35 | 105

OUTCOME MEASURES:

1. Primary Outcome: Procallagen-1 Amino-terminal Peptide (P1NP)
Time Frame: Baseline, Day 15, Day 30, Day 60, Day 90
Measure: Mean (Standard Error); unit: percentage change from baseline
Arm/Group | PTHrP 400 mcg/Day | PTHrP 600 mcg/Day | PTH 20 mcg/Day
Number analyzed (Participants) | 29 | 28 | 33
percentage change from baseline
  Day 15 | 32.54 (5.09) | 23.51 (7.04) | 60.67 (7.35)
  Day 30 | 48.89 (5.7) | 83.14 (12.48) | 97.27 (10.79)
  Day 60 | 34.71 (5.78) | 87.39 (22.24) | 125.46 (17.46)
  Day 90 | 46.07 (12.12) | 84.09 (20.57) | 171.49 (26.67)
Statistical Analysis 1: Comparison: PTHrP 400 mcg/Day vs PTHrP 600 mcg/Day vs PTH 20 mcg/Day; Test type: Non-Inferiority or Equivalence — An equivalence test of means for the percentage change in PINP and CTX using two one-sided tests applied to data from the parallel group design with a sample size of 31 in the PTH(1-34) group and 62 in the combined PTHrP(1-36) group achieved 80% power at 2.5% significant level for two-sided hypothesis testing (adjusted for the hypothesis testing at two key endpoints); p < 0.0005, Kruskal-Wallis — The reported p-value corresponds with percent change from baseline by day 15 in all three arms

2. Secondary Outcome: Changes in Bone Mineral Density of the Lumbar Spine.
Time Frame: 90 days
Measure: Mean (Standard Error); unit: Percent change from baseline
Arm/Group | PTHrP 400 mcg/Day | PTHrP 600 mcg/Day | PTH 20 mcg/Day
Number analyzed (Participants) | 29 | 28 | 33
Percent change from baseline | 1.89 (0.49) | 1.52 (0.61) | 2.17 (0.60)
Statistical Analysis 1: Comparison: PTHrP 400 mcg/Day vs PTHrP 600 mcg/Day vs PTH 20 mcg/Day; Test type: Non-Inferiority or Equivalence — Power calculations for this study were determined considering the expected effects of PTHrP (1-36) relative to PTH (1-34) on the primary endpoints of P1NP and CTX after 3 months of treatment relative to baseline using previously published data as weel as anticipated attrition rate. See primary outcomes; p < 0.05, Kruskal-Wallis — The reported p-value corresponds with percent change from baseline in all Arms/groups; The threshold for stasistical significance was p=0.05

3. Primary Outcome: Carboxy-terminal Telopeptides of Collagen-1 (CTX)
Time Frame: Baseline, Day 15, Day 30, Day 60, Day 90
Measure: Mean (Standard Error); unit: percentage change from baseline
Arm/Group | PTHrP 400 mcg/Day | PTHrP 600 mcg/Day | PTH 20 mcg/Day
Number analyzed (Participants) | 29 | 28 | 33
percentage change from baseline
  Day 15 | -12.40 (7.19) | 10.25 (10.66) | 4.87 (8.09)
  Day 30 | 1.60 (10.65) | 9.59 (16.49) | 13.89 (12.43)
  Day 60 | 4.13 (7.93) | 14.38 (15.89) | 52.98 (22.23)
  Day 90 | 32.65 (14.86) | 25.65 (11.75) | 92.46 (18.68)
Statistical Analysis 1: Comparison: PTHrP 400 mcg/Day vs PTHrP 600 mcg/Day vs PTH 20 mcg/Day; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p < 0.05, Kruskal-Wallis — The reported p-value corresponds with percent change from baseline at Day 60 and at Day 90 for the PTH group and at day 90 for the PTHrP 400 and PTHrP 600 groups

4. Secondary Outcome: Changes in Bone Mineral Density of the Total Hip.
Time Frame: 90 days
Measure: Mean (Standard Error); unit: Percent change from baseline
Arm/Group | PTHrP 400 mcg/Day | PTHrP 600 mcg/Day | PTH 20 mcg/Day
Number analyzed (Participants) | 29 | 28 | 33
Percent change from baseline | 0.68 (0.29) | 0.72 (0.30) | 0.54 (0.45)
Statistical Analysis 1: Comparison: PTHrP 400 mcg/Day vs PTHrP 600 mcg/Day vs PTH 20 mcg/Day; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p < 0.05, Kruskal-Wallis — The reported p-value corresponds with percent change from baseline in PTHrP 400 and 600 groups; The threshold for stastistical significance was p=0.05

5. Secondary Outcome: Changes in Bone Mineral Density of the Femoral Neck.
Time Frame: 90 days
Measure: Mean (Standard Error); unit: Percent change from baseline
Arm/Group | PTHrP 400 mcg/Day | PTHrP 600 mcg/Day | PTH 20 mcg/Day
Number analyzed (Participants) | 29 | 28 | 33
Percent change from baseline | 0.91 (0.41) | 0.54 (0.48) | 0.61 (0.49)
Statistical Analysis 1: Comparison: PTHrP 400 mcg/Day vs PTHrP 600 mcg/Day vs PTH 20 mcg/Day; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p < 0.05, Kruskal-Wallis — The reported p-value corresponds with percent change from baseline in the PTHrP 400 group; The threshold for stastistical significance was p=0.05

6. Secondary Outcome: Changes in Bone Mineral Density of the Forearm.
Time Frame: 90 days
Measure: Mean (Standard Error); unit: Percent change from baseline
Arm/Group | PTHrP 400 mcg/Day | PTHrP 600 mcg/Day | PTH 20 mcg/Day
Number analyzed (Participants) | 29 | 28 | 33
Percent change from baseline | -0.48 (0.61) | -0.99 (0.78) | -0.97 (0.49)
Statistical Analysis 1: Comparison: PTHrP 400 mcg/Day vs PTHrP 600 mcg/Day vs PTH 20 mcg/Day; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p > 0.05, Kruskal-Wallis — The reported p-value corresponds with percent change from baseline in all Arms/groups; The threshold for statistical signifcance was p=0.05

7. Secondary Outcome: Changes in Bone Mineral Density of the Distal 1/3 Radius.
Time Frame: 90 days
Measure: Mean (Standard Error); unit: Percent change from baseline
Arm/Group | PTHrP 400 mcg/Day | PTHrP 600 mcg/Day | PTH 20 mcg/Day
Number analyzed (Participants) | 29 | 28 | 33
Percent change from baseline | -0.35 (0.54) | -0.34 (0.96) | -0.82 (0.64)
Statistical Analysis 1: Comparison: PTHrP 400 mcg/Day vs PTHrP 600 mcg/Day vs PTH 20 mcg/Day; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p > 0.05, Kruskal-Wallis — The reported p-value corresponds with percent change from baseline in all Arms/groups; The threshold for statistical significance was p=0.05

8. Secondary Outcome: Total Serum Calcium (mg/dl)
Time Frame: Baseline, Day 15, Day 30, Day 60, Day 90
Measure: Mean (Standard Error); unit: mg/dl
Arm/Group | PTHrP 400 mcg/Day | PTHrP 600 mcg/Day | PTH 20 mcg/Day
Number analyzed (Participants) | 29 | 28 | 33
mg/dl
  Baseline | 9.48 (0.06) | 9.51 (0.06) | 9.49 (0.06)
  Day 15 | 9.95 (0.09) | 9.87 (0.09) | 9.57 (0.02)
  Day 30 | 9.73 (0.09) | 9.67 (0.06) | 9.55 (0.06)
  Day 60 | 9.71 (0.07) | 9.61 (0.06) | 9.58 (0.06)
  Day 90, time 0 | 9.56 (.07) | 9.45 (0.07) | 9.44 (0.06)
  Day 90, time 3 hours | 9.90 (0.08) | 9.76 (0.07) | 9.75 (0.06)
  day 90, time 6 hours | 9.90 (0.07) | 9.81 (0.10) | 9.78 (0.07)
Statistical Analysis 1: Comparison: PTHrP 400 mcg/Day vs PTHrP 600 mcg/Day vs PTH 20 mcg/Day; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p < 0.0005, F-test, one way analysis of variance — The reported p-value corresponds to change from baseline at Day 15 and 30 in the PTHrP 400 group and at Day 15 in the PTHrP 600 group; The threshold for statistical significance was p=0.05

9. Secondary Outcome: Serum Phosphorous
Time Frame: Baseline, Day 15, Day 30, Day 60, Day 90
Measure: Mean (Standard Error); unit: mg/dl
Arm/Group | PTHrP 400 mcg/Day | PTHrP 600 mcg/Day | PTH 20 mcg/Day
Number analyzed (Participants) | 29 | 28 | 33
mg/dl
  Baseline | 4.0 (0.07) | 3.93 (0.08) | 4.09 (0.08)
  Day 15 | 3.78 (0.07) | 3.68 (0.08) | 4.13 (0.08)
  Day 30 | 3.87 (0.09) | 3.71 (0.09) | 4.19 (0.11)
  Day 60 | 4.02 (0.07) | 3.97 (0.08) | 4.28 (0.08)
  Day 90 | 4.05 (0.09) | 3.98 (0.07) | 4.10 (0.07)
Statistical Analysis 1: Comparison: PTHrP 400 mcg/Day vs PTH 20 mcg/Day; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p < 0.05, F-test, one way analysis of variance — The reported p-value corresponds to PTH group on Day 60 compared to the PTHrP 400; The threshold for statistical significance was p=0.05
Statistical Analysis 2: Comparison: PTHrP 400 mcg/Day vs PTHrP 600 mcg/Day vs PTH 20 mcg/Day; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p < 0.005, Kruskal-Wallis — The reported p-value corresponds to the PTH group on Day 30 compared to the PTHrP 400 group and Day 60 compared to the PTHRp 600 group; The threshold for statistical significance was p=0.05
Statistical Analysis 3: Comparison: PTHrP 400 mcg/Day vs PTHrP 600 mcg/Day vs PTH 20 mcg/Day; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p < 0.0005, Kruskal-Wallis — The reported p-value correspond to the PTH group on Day 15 compared to the PTHrP 400 group and Day 15 and 30 compared to the PTHrP 600 group; The threshold for statistical significance was p=0.05

10. Secondary Outcome: 24 Hour Urine Calcium
Time Frame: 90 days
Measure: Mean (Standard Error); unit: mg/gm creatinine
Arm/Group | PTHrP 400 mcg/Day | PTHrP 600 mcg/Day | PTH 20 mcg/Day
Number analyzed (Participants) | 29 | 28 | 33
mg/gm creatinine
  Baseline | 206.37 (14.08) | 213.07 (16.22) | 209.99 (14.47)
  Day 90 | 260.46 (22.72) | 235.25 (20.34) | 232.48 (17.47)
Statistical Analysis 1: Comparison: PTHrP 400 mcg/Day vs PTHrP 600 mcg/Day vs PTH 20 mcg/Day; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p < 0.005, F-test, one way analysis of variance — The reported p-value corresponds to the increase from baseline to D90 in the PTHrP 400 group; the threshold for statistical significance was p=0.05

11. Secondary Outcome: 1,25 Vitamin D
Time Frame: Baseline, Day 15, Day 30, Day 60, Day 90
Measure: Mean (Standard Error); unit: pg/ml
Arm/Group | PTHrP 400 mcg/Day | PTHrP 600 mcg/Day | PTH 20 mcg/Day
Number analyzed (Participants) | 29 | 28 | 33
pg/ml
  Baseline | 49.06 (3.24) | 42.49 (2.20) | 42.51 (1.75)
  Day 15 | 84.92 (5.65) | 63.07 (4.71) | 65.25 (3.68)
  Day 30 | 76.04 (4.65) | 65.15 (3.71) | 67.29 (3.79)
  Day 60 | 67.85 (4.40) | 57.02 (4.07) | 58.15 (2.98)
  Day 90 | 64.36 (4.34) | 55.08 (4.20) | 53.73 (2.30)
Statistical Analysis 1: Comparison: PTHrP 400 mcg/Day vs PTHrP 600 mcg/Day vs PTH 20 mcg/Day; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p < 0.05, F-test, one way analysis of variance — The reported p value corresponds to an increased from baseline at all time points in all Arms/groups as well as to the increase in the in the PTHrP 400 group at Day 60 and 90 compared to the PTHrP 600 and PTH groups; the threshold for statistical significance was p=0.05
Statistical Analysis 2: Comparison: PTHrP 400 mcg/Day vs PTHrP 600 mcg/Day vs PTH 20 mcg/Day; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p < 0.005, Kruskal-Wallis — The reported p-value corresponds to the comparison of the PTHrP 400 group at Day 15 to the PTHrP 600 and PTH groups; The threshold for statistical significance was p=0.05

12. Secondary Outcome: Fractional Excretion of Calcium
Description: (Serum Creatinine X Urine Calcium)/(Serum Calcium X Urine Creatinine)
Time Frame: Baseline, Day 15, Day 30, Day 60, Day 90
Measure: Mean (Standard Error); unit: % excreted
Arm/Group | PTHrP 400 mcg/Day | PTHrP 600 mcg/Day | PTH 20 mcg/Day
Number analyzed (Participants) | 29 | 28 | 33
% excreted
  Baseline | 2.38 (0.21) | 2.71 (0.24) | 2.30 (0.23)
  Day 15 | 3.42 (033) | 4.18 (0.39) | 2.55 (0.27)
  Day 30 | 3.27 (0.34) | 3.74 (0.27) | 2.92 (0.34)
  Day 60 | 3.38 (0.34) | 2.89 (0.28) | 2.95 (0.29)
  Day 90 | 3.10 (0.25) | 2.89 (0.27) | 3.37 (0.37)
Statistical Analysis 1: Comparison: PTHrP 400 mcg/Day vs PTHrP 600 mcg/Day vs PTH 20 mcg/Day; Test type: Non-Inferiority or Equivalence — Power calculations for this study were determined considering the expected effects of PTHrP (1-36) relative to PTH (1-34) on the primary endpoints of P1NP and CTX after 3 months of treatment relative to baseline using previously published data as weel as anticipated attrition rate; p < 0.05, F-test, one way analysis of variance — The reported p-value corresponds to an increase compared to baseline in the PTHrP 600 group at D15 and D30; The threshold for stastistical significance was p=0.05
Statistical Analysis 2: Comparison: PTHrP 400 mcg/Day vs PTHrP 600 mcg/Day vs PTH 20 mcg/Day; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 12, analysis 1]; p < 0.005, Kruskal-Wallis — the reported p-value corresponds to change from baseline in the PTHrP 400 group at Day 15,30, 60 and 90 and the PTH group at day 90; the threshold for statistical significance was p=0.05

13. Secondary Outcome: Tubular Maximum for Phosphorous/Glomerular Filtration Rate (TMP/GFR)
Description: Fractional tubular reabsorption of phosphate (TRP) = 1-{(U phos/P phos) x ( P creat/U creat)} if TRP < or = 0.86 then TMP/GFR = TRP x P phos if TRP > 0.86 then TMP/GFR = 0.3 x TRP/{1-(0.8 x TRP)} x P phos
  U= urine, P = plasma
Time Frame: Baseline, Day 15, Day 30, Day 60, Day 90
Measure: Mean (Standard Error); unit: mg/dl
Arm/Group | PTHrP 400 mcg/Day | PTHrP 600 mcg/Day | PTH 20 mcg/Day
Number analyzed (Participants) | 29 | 28 | 33
mg/dl
  Baseline | 3.80 (0.11) | 3.71 (0.11) | 3.96 (0.12)
  Day 15 | 3.78 (0.14) | 3.47 (0.15) | 4.18 (0.12)
  Day 30 | 3.88 (0.14) | 3.61 (0.14) | 4.03 (0.12)
  Day 60 | 4.02 (0.14) | 3.84 (0.13) | 4.28 (0.13)
  Day 90 | 4.11 (0.11) | 3.90 (0.12) | 4.00 (0.13)
Statistical Analysis 1: Comparison: PTHrP 400 mcg/Day vs PTHrP 600 mcg/Day vs PTH 20 mcg/Day; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p < 0.05, Kruskal-Wallis — The reported p-value corresponds the PTH group on Day 15 compared to the PTHrP 400 group and to the PTHrP 600 group at Day 30 and Day 60; The threshold for statistical significance was p=0.05
Statistical Analysis 2: Comparison: PTHrP 600 mcg/Day vs PTH 20 mcg/Day; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 12, analysis 1]; p < 0.0005, Kruskal-Wallis — Thre reported p-value correspond to the PTH group compared to the PTHrp 600 group at day 15; the threshold for statistical significance was p=0.05

ADVERSE EVENTS:
Description: Adverse event data was collected at each study visit.
Arm/Group | PTHrP 400 mcg/Day | PTHrP 600 mcg/Day | PTH 20 mcg/Day
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/35 | 0/35
Other Adverse Events (participants affected / at risk) | 33/35 | 31/35 | 27/35
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PTHrP 400 mcg/Day (N=35) | PTHrP 600 mcg/Day (N=35) | PTH 20 mcg/Day (N=35)
Dermatologic (Skin and subcutaneous tissue disorders) | 19 | 23 | 14
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 7 | 8 | 10
Neurologic (Nervous system disorders) | 11 | 11 | 12
Psychological (Psychiatric disorders) | 5 | 11 | 12
Gastrointestinal (Gastrointestinal disorders) | 13 | 12 | 11
Infection (Infections and infestations) | 4 | 4 | 3
Cardiovascular (Cardiac disorders) | 0 | 4 | 2
Genitourinary (Renal and urinary disorders) | 3 | 0 | 2
Other (General disorders) | 17 | 15 | 20

LIMITATIONS AND CAVEATS:
This study was not double-blinded. There was no placebo group in this study. Subjects had higher than anticipated calcium intake and baseline vitamin D levels.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No